CLINICAL TRIAL: NCT02392637
Title: A Phase II Study of Gemcitabine, Cisplatin, and Abraxane in Advanced Biliary Cancers
Brief Title: Gemcitabine Hydrochloride, Cisplatin, and Nab-Paclitaxel in Treating Patients With Advanced or Metastatic Biliary Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0524; NCI-2015-00578 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0524 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Stage III Intrahepatic Cholangiocarcinoma AJCC v7; Stage IIIA Gallbladder Cancer AJCC v7; Stage IIIB Gallbladder Cancer AJCC v7; Stage IVA Gallbladder Cancer AJCC v7; Stage IVA Intrahepatic Cholangiocarcinoma AJCC v7; Stage IVB Gallbladder Cancer AJCC v7; Stage IVB Intrahepatic Cholangiocarcinoma AJCC v7; Unresectable Extrahepatic Bile Duct Carcinoma; Unresectable Gallbladder Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Treatment (nab-paclitaxel, cisplatin, gemcitabine) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel

SUMMARY:
This phase II trial studies how well gemcitabine hydrochloride, cisplatin, and nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation) work in treating patients with biliary cancers (which includes the gallbladder and bile ducts inside and outside the liver) that have spread to other places in the body and usually cannot be cured or controlled with treatment. Drugs used in chemotherapy, such as gemcitabine hydrochloride, cisplatin, and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the progression-free survival (PFS) of gemcitabine hydrochloride (gemcitabine), cisplatin, and nab-paclitaxel in advanced, untreated biliary cancers (intrahepatic cholangiocarcinomas, extrahepatic cholangiocarcinomas, and gallbladder cancers).

SECONDARY OBJECTIVES:

I. Determine the response rate (RR) and disease control rate (partial response + complete response + stable disease) of gemcitabine, cisplatin, and nab-paclitaxel in advanced biliary cancers.

II. Determine overall survival (OS) of gemcitabine, cisplatin, and nab-paclitaxel in advanced biliary cancers.

III. Evaluate the toxicity of gemcitabine, cisplatin, and nab-paclitaxel in advanced biliary cancers.

EXPLORATORY OBJECTIVES:

I. Correlate the carbohydrate antigen (CA) 19-9 response (defined as >50% decrease from baseline) with tumor response, PFS and OS.

II. Assess ribonucleotide reductase subunit MI (RRMI), excision repair cross-complementation group 1 (ERCC1) pre-treatment status and correlate with tumor response, PFS and OS on an exploratory basis.

III. Collect optional blood and tissue at the start of treatment and at progression to explore mechanisms of resistance.

OUTLINE:

Patients receive paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, or gallbladder cancer or may undergo a repeat biopsy for histologic confirmation if pre-existing biopsy is not sufficient for diagnosis
* Metastatic or unresectable disease documented on diagnostic imaging studies
* May not have received prior chemotherapy; if patient has received prior adjuvant therapy, must be > 6 months from treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Platelets >= 100,000/ul
* Hemoglobin > 9.0 g/dL
* Total bilirubin =< 1.5 mg/dL (in patients with known Gilbert's syndrome direct bilirubin =< 1.5 x upper limit of normal [ULN] will be used as organ function criteria, instead of total bilirubin)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) = < 5 x ULN
* Creatinine =< 1.5 gm/dL
* Negative serum or urine pregnancy test in women with childbearing potential (WOCBP) defined as not post-menopausal for 12 months or no previous surgical sterilization, within one week prior to initiation of treatment; WOCBP must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy
* A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy; if the partner is pregnant or breastfeeding, the subject must use a condom
* Patients must sign an informed consent and authorization indicating that they are aware of the investigational nature of this study and the known risks involved

Exclusion Criteria:

* Peripheral neuropathy of grade 2 or greater by Common Terminology Criteria for Adverse Events (CTCAE) 4.0; in CTCAE version 4.0 grade 2 sensory neuropathy is defined as "moderate symptoms; limiting instrumental activities of daily living (ADLs)"
* Concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study such as unstable angina, myocardial infarction within 6 months, unstable symptomatic arrhythmia, uncontrolled diabetes, serious active or uncontrolled infection
* Pregnancy (positive pregnancy test) or lactation
* Known central nervous system (CNS) disease, except for treated brain metastasis; treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]) during the screening period; anticonvulsants (stable dose) are allowed; treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, linear accelerator [LINAC], or equivalent) or a combination as deemed appropriate by the treating physician; patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to day 1 will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milind Javle, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Shroff RT, Javle MM, Xiao L, Kaseb AO, Varadhachary GR, Wolff RA, Raghav KPS, Iwasaki M, Masci P, Ramanathan RK, Ahn DH, Bekaii-Saab TS, Borad MJ. Gemcitabine, Cisplatin, and nab-Paclitaxel for the Treatment of Advanced Biliary Tract Cancers: A Phase 2 Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):824-830. doi: 10.1001/jamaoncol.2019.0270. PMID 30998813
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 2 clinical trial conducted at the University of Texas MD Anderson Cancer Center and the Mayo Clinic in Phoenix.
Pre-assignment Details: 62 participants enrolled, 60 started treatment and 2 did not receive treatment (1) Progressive disease and (1) Withdrew consent.
Groups:
- High Dosage: Gemcitabine 1000mg/m2, Cisplatin 25mg/m2 & Nab-Paclitaxel 125mg/m2 on days 1 & 8 of a 21 day cycle.
- Low Dosage: Gemcitabine 800mg/m2, Cisplatin 25mg/m2 & Nab-Paclitaxel 100mg/m2 on days 1 & 8 of a 21 day cycle.
Period: Overall Study
Arm/Group | High Dosage | Low Dosage
Started | 32 | 28
Completed | 32 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat participants
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dosage | Low Dosage | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Continuous [Median (Standard Deviation); unit: years] | 58.1 (11.1) | 58.8 (11.1) | 58.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 16 | 17 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 28 | 60
Tumor Type [Count of Participants; unit: Participants]
  Intrahepatic cholangiocarcinoma (IHCC) | 24 | 14 | 38
  Extrahepatic cholangiocarcinoma (EHCC) | 4 | 5 | 9
  Gallbladder Cancer (GBC) | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: up to 3 years
Population: 3 participants are not included due to 2 Discontinued during cycle 1 (adverse event) and 1 Refused treatment following cycle 1 (patient choice). The analysis for PFS were calculated for the total treated population that received both high and low dosage.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | High Dosage | Low Dosage
Number analyzed (Participants) | 31 | 26
months | 11.4 [6.0 to 15.6] | 14.9 [3.8 to NA] — Not estimable due to limited number of events
Statistical Analysis 1: Comparison: High Dosage vs Low Dosage; Test type: Superiority; p = 0.62, Log Rank

2. Secondary Outcome: Median Overall Survival (OS)
Description: The Kaplan-Meier method was used to estimate OS, with surviving patients censored at the time of surgery or at last known follow-up.
Time Frame: up to 3 years
Population: 3 participants are not included due to they were lost to follow up.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- High Dose: Gemcitabine 1000mg/m2, Cisplatin 25mg/m2 & Nab-Paclitaxel 125mg/m2 on days 1 & 8 of a 21 day cycle
- Low Dose: Gemcitabine 800mg/m2, Cisplatin 25mg/m2 & Nab-Paclitaxel 100mg/m2 on days 1 & 8 of a 21 day cycle.
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 31 | 26
months | 19.5 [10 to NA] — Not estimable due to limited number of events. | 15.7 [8.7 to NA] — Not estimable due to limited number of events.
Statistical Analysis 1: Comparison: High Dose vs Low Dose; Test type: Superiority; p = 0.39, Log Rank

3. Secondary Outcome: Number of Participants With Treatment Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria(RECIST v1.1.14) for target lesions and assessed by MRI: Complete Response (CR),Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 32 | 28
Participants
  Disease Control Rate(DCR) | 25 | 18
  Complete Response(CR) | 0 | 0
  Partial Response (PR) | 14 | 9
  Stable Disease(SD) | 11 | 9
  Progressive Disease(PD) | 3 | 5
  Unknown | 4 | 5

ADVERSE EVENTS:
Time Frame: up to 3 years
Arm/Group | High Dose | Low Dose
All-Cause Mortality (participants affected / at risk) | 1/32 | 0/28
Serious Adverse Events (participants affected / at risk) | 5/32 | 1/28
Other Adverse Events (participants affected / at risk) | 8/32 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=32) | Low Dose (N=28)
Neutropenia (Blood and lymphatic system disorders) | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=32) | Low Dose (N=28)
Neutropenia (Blood and lymphatic system disorders) | 8 | 9
Anemia (Blood and lymphatic system disorders) | 6 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 1
Elevated ALP (Blood and lymphatic system disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal Infection (Infections and infestations) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 1 | 0
Elevated AST (Blood and lymphatic system disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT02392637/Prot_SAP_000.pdf